CLINICAL TRIAL: NCT06577415
Title: A Single Dose Pharmacokinetic Study of ray1225 in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: A Study of RAY1225 in Participants With Impaired Liver Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1225-24-04
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment received single subcutaneous dose of 3 milligrams (mg) RAY1225.
  Interventions: Drug: RAY1225
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment received single subcutaneous dose of 3 mg RAY1225.
  Interventions: Drug: RAY1225
- Normal Hepatic Function (Active Comparator): Participants with normal hepatic function received single subcutaneous dose of 3 mg RAY1225.
  Interventions: Drug: RAY1225

INTERVENTIONS:
Drug: RAY1225 — Administered SC

SUMMARY:
The purpose of this study is to assess how fast RAY1225 gets into the blood stream and how long it takes the body to remove it in participants with impaired liver function compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 to ≤ 75 years;
2. BMI ≥ 20 kg/m2 up to ≤ 32 kg/m2;
3. Participants (including partners) must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product;
4. Signature of a dated Informed Consent Form (ICF) indicating that the participates has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment;
5. eGFR ≥ 60 mL/min/1.73 m2;

   Participants with Normal Hepatic Function Only:
6. Healthy males or females as determined by medical history, physical examination, and other screening procedures, with normal liver function;

   Participants with hepatic impairment only:
7. Males or females with chronic mild and moderate liver impairment, assessed by Child-Pugh scoring.

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product;
2. QTcF> 450ms;
3. Participants with serious infections, trauma, gastrointestinal surgery or other major surgical procedures within 4 weeks;
4. Participates who donated blood or bleeding profusely (> 400 mL) in the 3 months;
5. Pregnant or lactating women, or women of childbearing age with a positive pregnancy test;
6. Smoking averaged more than 10 cigarettes per day in the 3 months prior to screening;
7. Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2;

   Participants with Normal Hepatic Function Only:
8. Any history of hepatic impairment, or potential presence of liver function impairment by physical examination and laboratory examination at screening.

   Participants with Hepatic Impairment Only:
9. Any history of clinically serious illness or disease or condition except for primary liver disease that the investigator believes may affect the results of the trial, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, respiratory or hematological, immune, psychiatric, and metabolic disorders.
10. Participants with drug-induced liver injury; history of liver transplantation; cirrhosis in combination with the following complications: including but not limited to liver failure, hepatic encephalopathy, hepatocellular carcinoma, esophageal bleeding from ruptured fundic varices.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under The Drug Concentration-Time Curve From Zero To Infinity (AUC[0-∞]) of RAY1225 | DAY1~43
  Pharmacokinetics (PK): Area Under The Drug Concentration-Time Curve From Zero To Infinity (AUC[0-∞]) of RAY1225.
PK: Maximum Observed Drug Concentration (Cmax) of RAY1225 | DAY1~43
  PK: Maximum Observed Drug Concentration (Cmax) of RAY1225

SECONDARY OUTCOMES:
Number of participants with drug-related adverse events as assessed by CTCAE v5.0 | DAY1~43

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital,South Medical Hospital, Guangzhou, Guangdong, China